CLINICAL TRIAL: NCT05185037
Title: NIBP Algorithm Enhancements - MA_PM_NIBP Algorithm Enhancements_2021_11266
Brief Title: NIBP (Non-invasive Blood Pressure) Algorithm Enhancements (Characterize the Robustness of Motion Artifact Suppression)
Status: Terminated | Type: Observational
Why Stopped: Business decision with slower than expected enrollment..
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: MA_PM_NIBP_AE__2021_11266
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-06

CONDITIONS: Movement, Involuntary
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Caesarian Section Patient: Obstetric patient
  Interventions: Device: Philips IntelliVue X3 patient monitor with investigational NIBP measurement algorithm (measured once per 3 minutes)

INTERVENTIONS:
Device: Philips IntelliVue X3 patient monitor with investigational NIBP measurement algorithm (measured once per 3 minutes) — The purpose of this study is to compare measurements of NIBP taken by the study device and measurements taken by the current FDA-approved algorithm included in Rev. N.0 software for the IntelliVue patient monitors during motion artifact in patients undergoing caesarian section deliveries under epidural anesthesia

SUMMARY:
The study intervention consists of a non-invasive blood pressure (NIBP) measurement device and cuff (FDA-cleared Philips IntelliVue X3 Rev. N.04 patient monitor) running a non-approved modified software containing an enhanced measurement algorithm for NIBP.

DETAILED DESCRIPTION:
The purpose of this study is to compare measurements of NIBP taken by the study device and measurements taken by the current FDA-approved algorithm included in Rev. N.0 software for the IntelliVue patient monitors during motion artifact in patients undergoing caesarian section deliveries under epidural anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patient at Yale New Haven Hospital
* Receiving epidural anesthesia
* Age at least 18 years
* Willing and able to provide informed consent in a Sponsor approved language
* Willing and able to comply with study-related procedures
* Priority classification II, III, or IV

Exclusion Criteria:

* Non-caesarian section deliveries
* Ruptured uterus, prolonged fetal bradycardia, cord prolapse, or other emergent condition
* Procedures under general anesthesia
* Altered mental status
* Currently participating in another clinical trial with any product, treatment and/or medication that clinically interferes with the study endpoint(s)
* Priority classification I or V

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Laboring/Pregnant Females scheduled for Caesarean Section Delivery
Study Population: Pregnant Laboring Females scheduled for Caesarean Section Delivery
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
NIBP measurements with no technical alarms/INOPs | 1 Visit
  The primary endpoint for this study is the rate of NIBP measurements that are valid based on evaluation by a panel of three independent, licensed physicians. Valid measurement will include no technical alarm (INOP).
NIBP measurements with Diastolic, Systolic, and mean pressure within a physiologically plausible range for the patient population, treatment, and medication | 1 Visit
  The primary endpoint for this study is the rate of NIBP measurements that are valid based on evaluation by a panel of three independent, licensed physicians. Valid measurement will include Diastolic, Systolic, and mean pressures within a physiologically plausible range for the patient population, treatment and medication.
NIBP measurements with pulse pressure greater than 20% of the systolic blood pressure | 1 visit
  The primary endpoint for this study is the rate of NIBP measurements that are valid based on evaluation by a panel of three independent, licensed physicians. Valid measurement will include pulse pressure greater than 20% of the systolic blood pressure.

SECONDARY OUTCOMES:
Number of minutes between valid NIBP measurements compared to SoC | 1 visit
  The secondary endpoint for this study is the number of minutes between valid measurements for the investigational device as compared to the standard of care device.

CONTACTS AND LOCATIONS:
Overall Officials: Aymen Alian, MD, Principal Investigator — Yale New Haven Hospital
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Philips does not plan to share IPD data to other researchers.